CLINICAL TRIAL: NCT03650478
Title: Clinical Assessment of the NeuroBOX, a Cardio-respiratory Monitor Combined With a Fully Neurally Controlled Non-invasive Ventilator, in Infants.
Brief Title: Assessment of NeuroBOX and NeuroPAP in Infants.
Acronym: NeuroPap2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Maquet Critical Care (Unknown)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, Principal Investigator, Intensivist, Clinical Associate Professor, St. Justine's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUSJ-1841
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pediatric Respiratory Diseases; Bronchiolitis; Infant Respiratory Distress Syndrome
Keywords: Intensive Care; mechanical ventilation; noninvasive ventilation
MeSH Terms: conditions — Bronchiolitis; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Prospective single center crossover study with two different arms, one conducted in the Neonatal Intensive Care Unit and the other in the Pediatric Intensive Care Unit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premature infants group (Experimental): NeuroPAP ventilation (2h) and NeuroBox monitoring (23h)
  Interventions: Device: NeuroPAP ventilation (4h) and NeuroBox monitoring (25h)
- Bronchiolitis group (Experimental): NeuroPAP ventilation (4h) and NeuroBox monitoring (25h)
  Interventions: Device: NeuroPAP ventilation (2h) and NeuroBox monitoring (23h)

INTERVENTIONS:
Device: NeuroPAP ventilation (2h) and NeuroBox monitoring (23h) — Patients will be successively ventilated with conventional NIV (30 min with the conventional ventilator, 30 min with the NeuroBOX), and NeuroPAP (1 hour). An additional 20-hour period of recordings (with conventional NIV) will be conducted to characterize the neural breathing pattern, prevalence of apneas and tonic activation during conventional treatment. Finally, a second 1-hour period with NeuroPAP will be conducted
  Arms: Bronchiolitis group
Device: NeuroPAP ventilation (4h) and NeuroBox monitoring (25h) — Patients will be successively ventilated with conventional NIV (30 min with the conventional ventilator, 30 min with the NeuroBOX), and NeuroPAP (3 hours). An additional 20-hour period of recordings (with conventional NIV) will be conducted to characterize the neural breathing pattern, prevalence of apneas and tonic activation during conventional treatment. Finally, a second 1-hour period with NeuroPAP will be conducted
  Arms: Premature infants group

SUMMARY:
Non-invasive ventilation (NIV, delivered via a mask or cannulas) permits to reduce the need for tracheal intubation in infants who needs a ventilatory support. NIV can be delivered with nasal CPAP (continuous positive airway pressure) or NIPPV (nasal intermittent positive pressure ventilation). The synchronization of the respiratory support according to the patient's demand is very difficult to obtain in infants with the conventional ventilatory modes. In all these ventilatory modes, the end-expiratory pressure (PEEP) is fixed and set by the clinician. However, since infants are prone to alveolar collapse and must compensate for a non-compliant chest wall, an active and ongoing management of PEEP is very important to prevent the lung de-recruitment.

A new respiratory support system (NeuroPAP) has been developed to address these issues of synchronization and control of PEEP. This new system uses diaphragmatic tonic activity (Edi) that reflects the patient's efforts to increase lung recruitment and therefore it continuously controls the delivery of assist continuously both during inspiration (like NAVA) and during expiration, allowing a unique neural control of PEEP.

A new device, the NeuroBOX, permits to deliver NIV with NeuroPAP, CPAP, or NIPPV, and also to serve as a cardio-respiratory monitor, tracking and displaying cardiac and respiratory signals, trends, and cardio-vascular events.

The two main objectives of this study are: 1- To evaluate the clinical impact of NeuroPAP in infants with high tonic Edi; 2- To characterize the cardio-respiratory pattern and its relationship with cerebral perfusion of infants with noninvasive support, using the monitoring capacity of the NeuroBOX.

The investigators expect that NeuroPAP will permit to improve the efficiency of NIV in infants, through the better synchronization and the personalization of the expiratory pressure level in response to the patient needs.

This study will be conducted in two subgroups of patients at high risk of elevated tonic Edi and of cardio-respiratory events: a subgroup of premature infants and a subgroup of infants with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

For premature infants group:

* Preterm infants born at a gestational age (GA) between 25 weeks (+0/7 days) and 34 weeks inclusively
* With post-birth age : > 2 days (for birth GA >28 weeks) or > 6 days (GA <28weeks) and < 4 months
* on non-invasive support, including CPAP, NIPPV, or NAVA, with settings in the following range : Maximal inspiratory pressure (total, including PEEP) ≤ 20 cmH2O, and PEEP between 4 and 9 cmH2O, and FiO2 < 50%

For bronchiolitis group:

* Infants with a weight < 5kg and a clinical diagnosis of bronchiolitis.
* on non-invasive support, including CPAP, NIPPV, or NAVA with settings in the range: Delivered inspiratory pressure (total, including PEEP) ≤ 20 cmH2O and PEEP: 5-9 cmH2O, and FiO2 <60 %
* With persisting respiratory failure: presence of at least one of the following criteria:

  * Respiratory rate > 50 /min
  * Symptoms of respiratory distress: mWCAS > 3
  * FiO2 > 30% -
  * Inspiratory Edi consistently > 15 µV

Exclusion Criteria: for both premature infants and bronchiolitis groups

* Suspected or proven pneumothorax;
* Patient on high-flow nasal cannula or on NAVA;
* Contra-indications to the placement of a new nasogastric tube (e.g. severe coagulation disorder, malformation or recent surgery in cervical, nasopharyngeal or esophageal regions);
* Hemodynamic instability requiring inotropes;
* Severe respiratory instability requiring imminent intubation according to the attending physician, or FiO2 > 50% to achieve a SpO2>90%, or PaCO2 > 75 mmHg on the last blood gas;
* Patient for whom a limitation of life support treatments is discussed or decided;
* Refusal by the treating physician;
* Refusal by the parents or legal guardians.

Ages: 2 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in indices of respiratory unloading | Last 5-minute period of each condition phase
  The inspiratory and tonic Edi will be extracted from the NeuroBOX during each phase. The mWCAS, a clinical scale of work of breathing, will be blindly collected during each ventilatory condition in the bronchiolitis patients.
Incidence of cardio-respiratory events | over 25 hours (Entire recordings)
  the number of apneas >20s, with and without desaturations and with/without bradycardia, and the number of bradycardia will be extracted from the NeuroBOX. This is a descriptive analysis, not a comparative analysis.

SECONDARY OUTCOMES:
Change in End expiratory lung volume (EELV) level | 5-minute period before and after the change of ventilatory mode
  change in EELV will be assessed using the 3D video-derived volumetry, comparing the mean EELV level in the 5 minutes before and after the change of ventilatory mode (from conventional NIPPV to NeuroPAP and the reverse).
Change in Indices of cerebral oxygenation and perfusion | Last 5-minute period of each condition phase
  FDNIRS-DCS technology will be used to measure the indices of cerebral oxygen metabolism, blood flow and tissue hemoglobin saturation
Change in comfort level in preterm infants | Last 5-minute period of each condition phase
  assessed by the bedside nurse in charge using the Pain/Agitation component of the validated scale N-PASS (neonatal pain, agitation, and sedation scale). The Pain/Agitation component varies from 0 to 10, and a lower score reflects a better comfort.
Change in comfort level in infants with bronchiolitis. | Last 5-minute period of each condition phase
  assessed by the bedside nurse in charge using the validated scale FLACC (Face, Legs, Activity, Cry, Consolability scale). The FLACC score varies from 0 to 10 and a lower score reflects a better comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Emeriaud, MD PhD, Principal Investigator — CHU Sainte Justine, Université de Montréal
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No